CLINICAL TRIAL: NCT06672809
Title: Effects of Core Stability Training on the Function and Control of Deep Stabilizing Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungdong University (Other)
Responsible Party: Principal Investigator, Kyeongjin Lee, professor, Kyungdong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-05-013
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Core Stability
Keywords: Core Stability; Deep Stabilizing Muscles; Muscle Activation; Rehabilitation
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluators were blinded to the intervention details of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Stability Training Group (Experimental): This group receives core stability training aimed at strengthening deep stabilizing muscles, including the transversus abdominis, to improve lumbar support and control. Participants perform a 50-minute session three times per week over eight weeks, focusing on exercises using unstable surfaces like the Pilates reformer to enhance proprioception and core engagement.
  Interventions: Behavioral: Core Stability Training
- Control Group (Active Comparator): This group participates in aerobic exercise sessions as a comparative intervention. Participants engage in a 50-minute session three times per week over eight weeks. The exercise includes warm-up, a main session (walking at a controlled intensity), and cool-down, with intensity levels adjusted over time to match cardiovascular improvements.
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Core Stability Training — Participants in this group undergo core stability training sessions targeting deep stabilizing muscles. The exercises are designed to enhance spinal support and core control by activating the transversus abdominis and other core muscles. Sessions involve the use of a Pilates reformer and other unstable surfaces, fostering proprioceptive engagement and improved muscle coordination. Training is conducted three times per week for eight weeks, with each session lasting 50 minutes.
  Arms: Core Stability Training Group
Behavioral: Aerobic Exercise — Participants in this group engage in aerobic exercise sessions that consist of warm-up, controlled-intensity walking, and a cool-down phase. This intervention serves as a comparative baseline, aiming to improve cardiovascular endurance without specifically targeting core stability. The aerobic routine is adjusted over time to increase exercise intensity, conducted three times per week for eight weeks, with each session lasting 50 minutes.
  Arms: Control Group

SUMMARY:
This study investigates the effects of core stability training on the functionality and control of deep stabilizing muscles in healthy adults. Core stability exercises focus on strengthening the transversus abdominis and related core muscles to prevent and manage low back pain. Participants are randomly assigned to either the experimental group, performing core stability exercises on unstable surfaces such as a reformer, or the control group, performing aerobic exercises. Outcomes are measured by changes in muscle thickness and contraction time using rehabilitative ultrasound imaging, aiming to demonstrate the potential of core stabilization for enhancing spine support and reducing lower back pain.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 29 years
* Healthy adults who can understand and complete the planned training program
* Individuals who have signed informed consent to participate in the study

Exclusion Criteria:

* Individuals with balance disorders due to orthopedic or neurological conditions
* Those with cardiopulmonary diseases
* Individuals who have undergone surgery within the past 6 months
* Persons with other physical disabilities that could interfere with the study
* Individuals who have participated in similar studies recently
* Pregnant individuals

Ages: 20 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Thickness of Deep Stabilizing Muscles | Baseline and 8 weeks after the intervention
  The thickness of the core stabilizing muscles, including the rectus abdominis, transversus abdominis, internal oblique, and external oblique, is measured using rehabilitative ultrasound imaging (RUSI). For this assessment, a 10 MHz linear probe or a 3.5 MHz convex probe is positioned 2.5 cm lateral to the umbilicus while the participant lies in a supine position. The measurement captures the distance between the upper and lower fascial layers of each muscle, providing an indication of muscle thickness. Three measurements are taken, and the median value is used in analysis.
Contraction Time of Deep Stabilizing Muscles | Baseline and 8 weeks after the intervention
  This measure assesses the contraction time of deep stabilizing muscles, specifically during a hollowing exercise where the participant engages the transversus abdominis and other abdominal muscles. Using rehabilitative ultrasound imaging (RUSI), the probe is positioned 2.5 cm lateral to the umbilicus to observe muscle activation. Contraction time is recorded as the duration from the onset of muscle activation to full contraction. Measurements are taken three times, with the median value used for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, Kyungdong University, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No